CLINICAL TRIAL: NCT00214786
Title: Pancreatic Islet Cell Transplantation - A Novel Approach to Immunosuppression and Validation of Remote Site Islet Cell Processing, Islet Cell Culture and Two-Layer Preservation
Brief Title: Pancreatic Islet Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Baylor Health Care System (Other); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 003-040
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Mellitus; Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Hypoglycemia; Hyperglycemia | interventions — Islets of Langerhans Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Islet Cell Transplantation (Experimental): Allogenic islet cell transplantation
  Interventions: Biological: Islet cell transplantation

INTERVENTIONS:
Biological: Islet cell transplantation — Allogenic islet transplantation

SUMMARY:
The purpose of this study is to assess a novel approach to immunosuppression in allogenic pancreatic islet cell transplant recipients. In addition, the study aims to assess remote site islet processing with culture for pancreatic islet cell transplantation in human subjects.

DETAILED DESCRIPTION:
The purpose of this study is to assess a novel approach to immunosuppression in allogenic pancreatic islet cell transplant recipients. In addition, the study aims to assess remote site islet processing with culture for pancreatic islet cell transplantation in human subjects.

Detailed Description: Diabetes mellitus (DM) type I is a disease that has significant social and economical impact. The prevalence of the disease in the United States is about 120,000 in individuals aged 19 or less and 300,000 to 500,000 at all ages and 150 million worldwide.

So far there are no mechanical devices able to effectively adjust the dose of insulin injected according to the serum glucose in patients with DM. This leads to less than perfect sugar control, with episodes of hypoglycemia. Successful pancreas transplantation averts the need of insulin administration.

The emerging alternative to whole organ pancreas transplantation is pancreatic islet cell transplantation (ICT). The process is based on the enzymatic isolation of the pancreatic islets from an organ procured from a cadaver donor. The islets obtained are injected into the liver in the recipient via percutaneous catheterization of the portal venous system. This procedure allows the selective transplantation of the insulin-producing cell population avoiding open surgery as well as the transplantation of the duodenum and the exocrine pancreas and their related morbidity.

The initial efforts with ICT had only modest results. The immunosuppression regimen was similar to the one used in solid organ transplantation, based on high dose steroids and calcineurin inhibitors - both agents with diabetogenic effects. The results improved markedly with the changes in the manipulations of the islets, and the change in immunosuppression thus avoiding the higher doses of steroids and using sirolimus, tacrolimus and daclizumab initiated by the investigators group at the University of Alberta in Edmonton, Canada. Their protocol requires in general two islet cell infusions in order to attain the critical cell mass necessary to achieve insulin-independency. The changes in treatment were adopted as the Edmonton Protocol, which is used in several transplant centers, worldwide.

A novel approach to organ preservation uses the two-layer preservation technique. This allows for longer travel time for the eventual shipment of the pancreas to an islet cell processing facility remotely located from the donor procurement site.

The isolation of the islets from the donor pancreas will be performed at the Diabetes Research Institute in Miami, Florida, according to the standard currently used by that institution. The Diabetes Research Institute is a well-established center with a state-of-the-art islet cell isolation facility for the purpose of transplantation in humans, accredited and monitored by the FDA according to FDA standards.

The focus of the research in the ICT is centered on the development of a safe and effective procedure that will eventually replace surgical pancreas transplantation together with an ideal immunosuppressive regimen that provides safe and effective prevention against rejection, while minimizing the adverse events associated that negatively impact transplant recipient's quality of life.

This study is being conducted as a validation of the Edmonton protocol for ICT at our institution. Our aim is to test the efficacy of the use of the two-layer preservation technique for transport of the donor pancreas to the off-site processing facility and the use of islet cell culture in the off-site processing facility before the islet isolate is shipped to our center.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been fully informed and has signed an Institutional Review Board (IRB) approved informed consent form and is willing and able to follow study procedures for the full 2 years
2. Patient is expected to receive an islet cell transplant (up to 3 infusions) for type I diabetes mellitus

   * Type I diabetes of more than 5 years duration
   * Age between 18 and 65
   * Unstable diabetes mellitus control, as defined by glucose measurements above 200 mg/dL and/or below 80 mg/dL despite adequate medical care
   * Hypoglycemia unawareness, as defined by episodes of loss of cognitive function
   * Incapacitating signs and symptoms, as defined by the referring physician
   * Poor control of HbA1c > 8%
   * Psychogenically able to comply, in the opinion of the investigator
3. Female patients of childbearing potential must have a negative urine or serum pregnancy test upon hospitalization or within 7 days prior to enrollment and have agreed to utilize effective birth control throughout the study as well as for 6 weeks following study completion.

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from study participation.

1. Patient has previously received or is receiving an organ or bone marrow transplant
2. Patient has a known hypersensitivity to Tacrolimus, sirolimus, daclizumab, or CellCept
3. Patient is pregnant or lactating
4. Patient has participated in a blinded trial or participated in a trial involving a non-marketed (investigational) drug within 3 months of enrollment
5. Patient has participated in a trial involving a marketed drug or an infusion device within 30 days of the start of the trial
6. Glomerular filtration rate (GLOFIL) < 60 mL/min
7. Serum Creatinine > 1.6 mg/dL consistently
8. Body mass index > 30
9. Autoimmune thyroiditis
10. Malignancy other than basal cell carcinoma or squamous cell carcinoma
11. Radiographic evidence of pulmonary infection
12. Evidence of liver disease
13. Portal hypertension
14. Active infections
15. Hypercoagulable states (history of recurrent venous thrombosis, defined thrombophilia)
16. Bleeding / coagulation disorders
17. Basal insulin C-Peptide > 0.3 ng/dL
18. Insulin C-peptide > 0.3 ng/dL during stimulation test
19. HbA1c > 12%
20. Insulin requirement > 1 IU/kg/day
21. Seropositivity for Human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV), Human T-cell leukemia virus-1 (HTLV-1)
22. Abnormal Pap smear in the last two months, active gynecological infection
23. Positive exercise or chemical tolerance test
24. Steroid dependence
25. Substance/alcohol abuse
26. Untreated proliferating diabetic retinopathy aa) Purified protein derivative (PPD) conversion or positive PPD without isonicotinic acid hydrazide (INH) bb) No Primary care physician or primary care physician less than 6 months cc) Smoking in the last 6 months dd) Abnormal Complete Blood Count (CBC) / Hemoglobin < 12 g/dL ee) Macroalbuminuria > 300 mg/24 hours ff) History of thyroid disease other than autoimmune disease gg) Untreated hyperlipidemia - Total Cholesterol (TC) > 240 mg/dL, Triglycerides (TGC) > 200 mg/dL, Low Density Lipoprotein (LDL) > 140 mg/dL hh) Untreated hyponatremia, hypokalemia, hypercalcemia, hypocalcemia ii) Iodine contrast allergy jj) Prostate Specific Antigen (PSA) > 4 kk) Panel Reactive Antibody (PRA) > 20% ll) Active peptic ulcer disease/gallstones/hemangioma mm) Abnormal mammogram

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2005-04; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlon Levy, MD, Principal Investigator — Baylor Regional Transplant Institute
Locations (1):
- Baylor Regional Transplant Institute - Baylor University Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period took place between April 2003 thru November 2005. Consent took place in the transplant clinic at Baylor University Medical Center (BUMC).
Pre-assignment Details: Patients signed informed consent after a consultation visit with tyhe PI. Then they proceeded through the evaluation phase of the study. During this phase, some patients were excluded based off of clinical findings (i.e. lab reports or procedures that did not meet protocol standards).
Groups:
- Islet Cell Transplantation: Patients who received islet cell transplantation. The recipients will be given islet cell preparation with more than 4000 Islet Equivalent (IE)/kg for multiple times up to 3 infusions.
Period: Overall Study
Arm/Group | Islet Cell Transplantation
Started | 4
Completed | 1
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Islet Cell: Patients with allogeneic islet cell transplantation
Arm/Group | Islet Cell
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (11.56143)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Achievement of Insulin Independence at 12-month Post Transplant
Description: To assess the number of patients who achieve insulin independence at 12-month after islet cell transplantation
Time Frame: 12 months post transplant
Measure: Number; unit: participant
Groups:
- Islet Cell: Allogeneic Islet Cell Transplantation
Arm/Group | Islet Cell
Number analyzed (Participants) | 4
participant | 1

2. Secondary Outcome: Presence or Absence of Hypoglycemic Unawareness
Description: Number of patients who achieved absence of hypoglycemic unawareness
Time Frame: 12 months after transplantation
Measure: Number; unit: participants
Arm/Group | Islet Cell
Number analyzed (Participants) | 4
participants | 3

3. Secondary Outcome: Incidence of Hypoglycemic Episodes
Description: Blood glucose <70 mg/dl, number of times reported per month
Time Frame: 12 months after transplantation
Measure: Mean (Standard Error); unit: episodes per month
Arm/Group | Islet Cell
Number analyzed (Participants) | 4
episodes per month | 7.3 (2.5)

4. Secondary Outcome: Change of Insulin Requirements in Patients Who Did Not Become Insulin Independent
Description: Percentage of insulin requirement at month 12 against that at baseline in the patients who did not achieve insulin independence. The percentage less than 100% indicates that subjects reduced insulin requirements 12 months after islet transplantation when compared with those at pre-transplant, while the parentage more than 100% represents that patients needed higher amount of exogenous insulin 12 months after islet transplantation.
Time Frame: 12 months after transplantation
Measure: Mean (Standard Error); unit: Percent decrease compared to baseline
Arm/Group | Islet Cell
Number analyzed (Participants) | 3
Percent decrease compared to baseline | 34.3 (10.5)

5. Secondary Outcome: Islet Cell Mass Obtained After Remote Site Processing
Description: The sum of Islet mass obtained after transport using the two-layer preservation method, remote site processing and islet culture. Islet mass as defined by Islet Equivalent per kilogram recipient body weight.
Time Frame: At transplantation
Measure: Mean (Standard Error); unit: Islet Equivalent per kilogram
Arm/Group | Islet Cell
Number analyzed (Participants) | 4
Islet Equivalent per kilogram | 8717 (2243)

6. Secondary Outcome: The Number of Islet Cell Infusions Needed to Achieve Insulin Independence
Time Frame: 12 months after transplantation
Measure: Mean (Standard Error); unit: number of infusion
Arm/Group | Islet Cell
Number analyzed (Participants) | 1
number of infusion | 2 (0)

7. Secondary Outcome: Renal Function
Description: Glomerular filtration rate measured by sodium iothalamate I-125 injection (GLOFIL)
Time Frame: 12 months after transplantation
Measure: Mean (Standard Error); unit: ml/min
Arm/Group | Islet Cell
Number analyzed (Participants) | 4
ml/min | 127.3 (7.9)

8. Secondary Outcome: Morbidity Related to the Immunosuppression Regimen
Description: Number of participants who experienced serious adverse events related to immunosuppression regimen
Time Frame: 12 months after transplantation
Measure: Number; unit: participant
Arm/Group | Islet Cell
Number analyzed (Participants) | 4
participant | 2

9. Secondary Outcome: Morbidity Related to the Islet Cell Infusion
Description: Number of participants who experienced serious adverse events related to islet cell infusion
Time Frame: 12months after transplantation
Measure: Number; unit: participant
Arm/Group | Islet Cell
Number analyzed (Participants) | 4
participant | 3

10. Secondary Outcome: The Quality of Life of the Recipients Measured With the RAND 36-item Short Form Health Survey
Description: Averaged score in subscales of 'physical functioning', 'Role limitations due to emotional problems', 'energy/fatigue', 'emotional well-being', 'social functioning', 'pain' and 'general health' in the RAND 36-item short form health survey (SF-36). Full scale range is 0-100 for all subscales with 100 as the best outcome and 0 as the worst outcome.
Time Frame: 12 months after transplantation
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Islet Cell
Number analyzed (Participants) | 4
Scores on a scale | 79.6 (12.4) [57.8 to 88.8]

ADVERSE EVENTS:
Time Frame: 12 months after transplantation
Description: The number of adverse events which was observed within 12 months after transplantation
Arm/Group | Islet Cell
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Cell (N=4)
Elevated Liver Function Tests (Hepatobiliary disorders) | 4 (4) — Three patients had elevated liver function tests post transplant and 1 patient had gallbladder hemorrhage.
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) — Patient experienced N & V which the PI determined was related to the protocol stated immunosuppressive medications.
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Islet Cell (N=4)
mouth ulcer (Skin and subcutaneous tissue disorders) | 4 (4)
nausea and vomiting (Gastrointestinal disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Three of the four patients voluntarily withdrew from the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No